CLINICAL TRIAL: NCT07106866
Title: A Comparative Evaluation of Double Versus Loop Suture Techniques in Sacrospinous Ligament Fixation Over Two Years
Brief Title: LOOP VS DOUBLE SUTURE TECHNIQUES IN SACROSPINOUS FIXATION: A TWO-YEAR STUDY
Status: Completed | Type: Observational
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ayse Betul Albayrak Denizli, MD, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: SSFtecnique
Record Dates: First submitted 2025-07-03; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Organ Prolapse; Surgical Procedure; Complications, Late Effect of Complications
Keywords: urogynecology; pelvic organ prolapse; sacrospinous ligament fixation; prolapse recurrence
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Double Suture Technique: Double Suture Technique - classical SSF using two individual permanent sutures.
  Interventions: Procedure: sacrospinous ligament fixation
- Loop Suture Technique: Loop Suture Technique - SSF using a single loop-style suture
  Interventions: Procedure: sacrospinous ligament fixation

INTERVENTIONS:
Procedure: sacrospinous ligament fixation — A longitudinal incision was made at the midline of the posterior vaginal wall, extending approximately 2-3 cm from the perineal body to the vaginal apex to form a tunnel. The incised vaginal epithelium was dissected from the underlying muscularis layer. Dissection was continued to the level of the ischial spine. The rectum was medialized to access the perirectal space. Upon palpating the ischial spine, the sacrospinous ligament was identified medial to it. Long retractors were placed over the ischial spine to protect the pudendal neurovascular structures. The bladder was retracted superiorly, and the rectum medially, for optimal visualization. Two separate or a loop 1-0 polypropylene suture(s) were placed approximately 1.5 fingerbreadths medial to the ischial spine on the ligament using a needle holder. These sutures were passed through the posterior vaginal tunnel to the apex and tied to secure the vaginal apex to the ligament

SUMMARY:
This retrospective cohort study aimed to compare clinical outcomes between the classical double suture technique and a modified loop suture technique used in sacrospinous ligament fixation for stage 3 or 4 pelvic organ prolapse. A total of 195 patients underwent surgery at a tertiary care center between January 2020 and January 2023. The primary outcome was the rate of reoperation due to recurrence within 24 months. Secondary outcomes included operative time, prolapse recurrence rate, and postoperative complications such as gluteal pain. The study was designed to evaluate whether a simplified suture method could improve surgical efficiency and patient recovery without compromising anatomical success.

DETAILED DESCRIPTION:
Sacrospinous ligament fixation is a commonly used surgical procedure for apical pelvic organ prolapse, particularly in women with advanced-stage prolapse who desire a native tissue repair approach. With increasing concerns regarding mesh-related complications, sacrospinous fixation has regained popularity as a mesh-free alternative.

This retrospective cohort study was conducted to evaluate and compare the clinical performance of two different suture techniques: the classical double suture method and a modified loop suture method. The main objective was to assess whether the loop suture technique, which involves a single point of tension, offers advantages in terms of operative efficiency and patient outcomes.

A total of 195 patients with stage 3 or 4 pelvic organ prolapse underwent sacrospinous ligament fixation between January 2020 and January 2023 at a tertiary urogynecology center. One group received the standard double suture technique, while the other underwent fixation using a single loop suture. All surgeries were performed by the same experienced surgical team.

The primary outcome was reoperation rate due to recurrence within 24 months. Secondary outcomes included total operative time, recurrence rate (as defined by POP-Q stage ≥2), and postoperative complications such as gluteal pain and rectal injury.

This study aims to provide evidence on whether a technical modification in a widely accepted native tissue repair procedure can improve surgical safety and reduce long-term complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 or 4 apical pelvic organ prolapse
* Underwent SSF between Jan 2020 and Jan 2023

Exclusion Criteria:

* Concomitant malignancy
* Previous apical prolapse surgery

Ages: 30 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — As uterine prolapse occures only in women
Study Population: Women aged 30 to 80 years with stage 3 or 4 apical pelvic organ prolapse who underwent sacrospinous ligament fixation at a tertiary urogynecology center. All patients were treated between January 2020 and January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Reoperation rate | 24 months
  Reoperation rate due to prolapse recurrence within 24 months

SECONDARY OUTCOMES:
Total operative time (in minutes) | up to 200 minutes
Postoperative complications (e.g. gluteal pain, hematoma) | 24 months
Prolapse recurrence rate (Stage ≥2 on POP-Q) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Women and Children's Diseases Training and Research Hospital, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided